CLINICAL TRIAL: NCT00717483
Title: BMI and Its Relationship to Hypoglycemic Seizures in Children With Insulin-requiring Diabetes
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rubina Heptulla, MD, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-23285
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 1 diabetes: children with type 1 diabetes

SUMMARY:
The landmark study Diabetes Control and Complication Trial (DCCT) clearly showed that intensive insulin management delays the onset and progression of longterm complications in adolescents with type 1 diabetes mellitus (T1DM). The same clinic trial also showed increased rate of severe hypoglycemia which required assistance. The risks of severe hypoglycemia, defined as loss of consciousness or seizure associated with hypoglycemia, include lower HbA1C, younger age, higher insulin dose, male sex, lower parental socioeconomic status, non-Hispanic white ethnicity, longer duration of disease, the presence of psychiatric disorders, and underinsurance.

The purpose of this protocol is to explore the relationship between hypoglycemic seizures and BMI.

DETAILED DESCRIPTION:
This is a retrospective study using questionnaire/survey/interview. We will give subjects a letter stating the purpose and describing the study. We will answer all questions they have about the study. Once the parents and patient verbally agree to participate in the study, we will proceed with the survey.

ELIGIBILITY:
Inclusion Criteria:

* T1DM
* 2-17 years old

Exclusion Criteria:

* T2DM
* Known seizure disorder

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects are patients with type 1 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubina A Heptulla, MD, Principal Investigator — Baylor (now Montefiore)
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Texas Childrens Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Effect of intensive diabetes treatment on the development and progression of long-term complications in adolescents with insulin-dependent diabetes mellitus: Diabetes Control and Complications Trial. Diabetes Control and Complications Trial Research Group. J Pediatr. 1994 Aug;125(2):177-88. doi: 10.1016/s0022-3476(94)70190-3. PMID 8040759
- [Background] Hypoglycemia in the Diabetes Control and Complications Trial. The Diabetes Control and Complications Trial Research Group. Diabetes. 1997 Feb;46(2):271-86. PMID 9000705
- [Background] Bulsara MK, Holman CD, Davis EA, Jones TW. The impact of a decade of changing treatment on rates of severe hypoglycemia in a population-based cohort of children with type 1 diabetes. Diabetes Care. 2004 Oct;27(10):2293-8. doi: 10.2337/diacare.27.10.2293. PMID 15451890
- [Background] Rewers A, Chase HP, Mackenzie T, Walravens P, Roback M, Rewers M, Hamman RF, Klingensmith G. Predictors of acute complications in children with type 1 diabetes. JAMA. 2002 May 15;287(19):2511-8. doi: 10.1001/jama.287.19.2511. PMID 12020331